CLINICAL TRIAL: NCT06727825
Title: Evaluation of Grass Pollen Sensitization Among Professionals Exposed or Not Exposed to Flour
Acronym: GRAMIPRO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: GRAMIPRO
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma; Sensitization
Keywords: Wheat flour; Occupational asthma; Grasses
MeSH Terms: conditions — Asthma; Asthma, Occupational

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Occupational asthma are a major etiology of allergic asthma, especially among manual labor. The baker job exposes to significant level of flour. Some of allergenic components at work have simitudes with environmental allergens, for example cereals flour with gramineous pollens.

GRAMIPRO is a retrospective cohort study that analyzes data from one specialized center at Créteil in the Paris region. The primary goal is to assess Participants include women and men aged over 18 years old at the time of their first consultation in the Occupational and Environmental Pathology Department of Créteil between April 2011 and July 2023, in order to explore asthma from an allergological perspective, patients working as bakers, pastry chefs, or restaurant workers, who are aware of exposed and patients in other professions; asthmatic patients with or without associated rhinitis.

Exclusions apply for patients who opposing to participate, patients without asthma symptoms; and patients who did not consult for the first time in the given period.

Data will be stored, anonymized, and analyzed using EasyMedStat. Data collection is scheduled between January 1 and 31, 2025 This research aims to o explore the factors that may influence the occurrence and severity of flour-induced allergic asthma symptoms in professionals exposed to this allergen, in order to consider prevention strategies and tools to advise individuals pursuing careers that expose them to flour. This study is intended for allergists, occupational physicians, general practitioners, and pulmonologists.

DETAILED DESCRIPTION:
15% of adult asthma cases are related to occupational exposure. Bakers are among the professions at the highest risk of developing allergies, particularly respiratory allergies. Cereals, including flour, are identified as a major cause. Cereals belong to the Poaceae family (wheat, rice, corn, barley, oats, rye, millet…). They are grasses, which gives them cross-allergenicity with grass pollens that are Group 4 allergens (83% homology between Phl p 4 and cereals). However, the professional factors and predispositions that might influence the occurrence and severity of asthma are not known. This study proposes, through an analysis of various data collected from bakers who consulted over a period of more than 10 years for asthma-related issues, as well as a comparison to other populations of workers who also consulted for asthma issues, to explore potential factors that seem relevant to investigate in more detail in the future.

GRAMIPRO is a retrospective cohort study that analyzes data from one Parisian center specialized in occupational dermatology and allergology - Centre Hospitalier Intercommunal de Créteil. This center is recognized at the national level as the Occupational and Environmental Disease Consultation Center (Centre de Consultation de Pathologies Professionnelles et de l'Environnement).

The primary goal is to analyze the impact of the prevalence of pollen grass sensitization in professionals with asthma, whether or not associated with allergic rhinitis, and exposed to flour or other allergens besides flour.

Secondary objectives focuses on the onset time and severity of respiratory symptoms (rhinitis and asthma) between patients sensitized and not sensitized to grass pollen by comparing FEV1 (in absolute and theoretical values), the FEV1/VC ratio, and the expected number of years from the onset of the first symptoms to the date of the first consultation The Inclusion criteria require to be aged 18 or older at the date of the first consultation. Further criteria are to have consulted for asthma-allergology related motifs between Patient identification involves querying the National Network for Surveillance and Prevention of Occupational Diseases (RNV3P, Réseau National de Vigilance et de Prévention des Pathologies professionnelles). Eligible patients will be informed by mail or post, and if no opposition expressed, their data will be collected and stored anonymously for analysis. Patient data will be collected from medical records, anonymized, and stored securely. Data collection is programmed between January 1 and 31, 2025. The study comprises patients from one center. In total, 405 patients were included, consisting of 135 cases and 2 matched controls for each case based on age, gender, date of first consultation, and type of tests conducted.

The collected data will include:

Initials of last name and first name, month and year of birth, sex, age on the day of consultation Referral type between occupational physician, general practitioner and specialist.

Start date of the profession Date of first consultation Presence of confirmed nasosinusis polyposis Date of symptom onset Smoking habits and status Maintenance and rescue treatments for asthma Hospitalization caused by an asthma attack Symptoms of rhinitis, asthma and conjunctivitis, Atopic history: asthma, atopic dermatitis, rhinitis, food and medication allergy, COPD Other known allergies: dust mites, mold, animal dander, tree and grass pollen… PFT: FEV1, Tiffeneau index, reversibility, Methacholine, PTN Prick Tests, Pulmonary Function Testing, biological analyzes Social security scheme: employee/self-employed Activity sector (NAF Code) Job position (CITP-8 Code) Work environment including : artisanal/industrial flour, hood, cleaning frequency, ventilation, individual protection Socio-professionnal outcome such as Recognition as an occupational disease and professional retraining Occupationnal specific IgE and this relative to grass pollen

Statistical analyses will use EasyMedStat to respond to the primary and secondary objectives.

The study has been officially approved by the Local Ethics Committee (CEL) of Créteil on the July 10th, 2024.

In conclusion, this research aims to explore predisposing factors in flour-induced allergic asthma to enable the implementation of individual and collective respiratory preventive measures in the workplace. Based on the results obtained, the study will allow the adaptation of preventive messages to be transmitted early to young atopic individuals sensitized to grass pollens who have a professional project exposing them to flour.

ELIGIBILITY:
Inclusion Criteria:

* patients who consulted between April 2011 and July 2023 for an occupational asthma
* active subjects
* Over 18 years at the first consultation with no upper limit
* Having not expressed their opposition to participate in the study

Exclusion Criteria:

* patients who opposing to participate in study
* patients without asthma symptoms
* patients who did not consult for the first time in the given period.
* Patient without occupational activity the day of the first consult or in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consulted between April 2011 and July 2023 for an occupational asthma exposed to flour or not at work
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
impact of the prevalence of pollen grass sensitization in professionals with asthma, whether or not associated with allergic rhinitis, and exposed to flour or other allergens besides flour. | Day1

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France